CLINICAL TRIAL: NCT00279760
Title: A Pilot, Multi-Center, Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Safety, Preliminary Clinical Activity and Immunogenicity of Multiple Doses of LEA29Y and CTLA4Ig Administered Intravenously to Subjects With Rheumatoid Arthritis
Brief Title: Phase I/II Multiple-Dose LEA29Y vs CTLAG4Ig vs Placebo in Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM103-002
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

INTERVENTIONS:
Drug: Belatacept
Drug: Abatacept

SUMMARY:
This randomized, double-blind, placebo controlled, parallel and multiple dose study provided safety, preliminary efficacy, and immunogenicity information about the use of BMS-188667 and BMS-224818 in subjects with RA

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA < 5 years
* Functional class I, II, or II as defined by the American College of Rheumatology (ACR) criteria.
* Must have failed at least 1 Disease Modifying Anit-Rheumatic Drug (DMARD)
* Joint count of 10 or more swollen and 12 or more tender.
* Erythrocyte Sedimentation Rate (ESR) > - 28mm/rr or norning stiffness > - 45 minutes.

Exclusion Criteria:

* Women and men who are not willing to use an accepted form of contraception.
* Active vasculitis
* Treatment with another investigational drug within 30 days
* History of asthma, angioedema, or anaphylaxix

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210
Dates: Primary Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
Assess the relative safety and preliminary efficacy (clinical activity) of BMS-188667 and BMS-224818 in subjects with rheumatoid arthritis (RA)

SECONDARY OUTCOMES:
Assess the immunogenicity of BMS-188667 and BMS-224818 in subjects with RA, and in a site specific substudy to the protocol, the pharmacokinetics (PK) and pharmacodynamics (PD) of BMS-188667 and BMS-224818 in subjects with RA

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (60):
- United States (20):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Huntsville, Alabama
  - Local Institution, Phoenix, Arizona
  - Local Institution, Tucson, Arizona
  - Local Institution, Los Angeles, California
  - Local Institution, San Diego, California
  - Local Institution, Miami, Florida
  - Local Institution, Chicago, Illinois
  - Local Institution, Boston, Massachusetts
  - Local Institution, Duluth, Minnesota
  - Local Institution, New Brunswick, New Jersey
  - Local Institution, New York, New York
  - Local Institution, Chapel Hill, North Carolina
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Cleveland, Ohio
  - Local Institution, Portland, Oregon
  - Local Institution, Nashville, Tennessee
  - Local Institution, Dallas, Texas
  - Local Institution, Salt Lake City, Utah
  - Local Institution, Seattle, Washington
- Belgium (6):
  - Local Instiution, Brussels
  - Local Institution, Diepenbeek
  - Local Institution, Ghent
  - Local Institution, Liège
  - Local Institution, Mons
  - Local Institution, Pellenberg
- Canada (9):
  - Local Institution, Edmonton, Alberta
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Calgary, Ontario
  - Local Institution, Ottawa, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
  - Local Institution, Sherbrook, Quebec
  - Local Institution, Ste-Foy, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- France (7):
  - Local Institution, Lille
  - Local Institution, Lyon
  - Local Institution, Montpellier
  - Local Institution, Paris
  - Local Institution, Rennes
  - Local Institution, Strasbourg
  - Local Institution, Toulouse
- Germany (9):
  - Local Institution, Berlin
  - Local Institution, Düsseldorf
  - Local Institution, Erlangen
  - Local Institution, Fankfurt
  - Local Institution, Hanover
  - Local Institution, Leipzig
  - Local Institution, München
  - Local Institution, Münster
  - Local Institution, Ratingen
- Ireland (2):
  - Local Institution, Cork
  - Local Institution, Dublin
- Netherlands (3):
  - Local Institution, Amsterdam
  - Local Institution, Leiden
  - Local Institution, Nijmegen
- Local Institution, Bern, Switzerland
- United Kingdom (3):
  - Local Institution, Birmingham
  - Local Institution, Cambridge
  - Local Institution, Leeds